CLINICAL TRIAL: NCT02154646
Title: A Phase 1b Study of LY2157299 in Combination With Gemcitabine in Patients With Advanced or Metastatic Unresectable Pancreatic Cancer
Brief Title: A Study of LY2157299 in Participants With Pancreatic Cancer That is Advanced or Has Spread to Another Part of the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14855; H9H-JE-JBAO (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-05-14; First posted 2014-06-03 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — LY-2157299; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LY2157299 + Gemcitabine (Experimental): 150 mg LY2157299 is administered orally twice daily for 14 days followed by 14 days without study drug (28 day cycle.) Gemcitabine 1000 milligram per square meter will be administered intravenously (IV) on Days 8, 15, and 22 in each cycle (28 day cycle). Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: LY2157299; Drug: Gemcitabine

INTERVENTIONS:
Drug: LY2157299 — Administered orally
Drug: Gemcitabine — Administered IV

SUMMARY:
The main purpose of this study is to evaluate the safety and side effects of LY2157299 in combination with gemcitabine in Japanese participants with pancreatic cancer that is advanced or has spread to another part of the body.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological diagnosis of adenocarcinoma of the pancreas that is locally advanced or metastatic and not amenable to resection with curative intent. These participants may have received prior chemotherapy, radiotherapy, cancer-related hormone therapy, or other investigational therapy as treatment or chemotherapy.
* Participants with previous radical surgery for pancreatic cancer are eligible after progression is documented.
* Have measurable disease or non-measurable disease, defined according to Response Evaluation Criteria in Solid Tumors (RECIST).
* Have given written informed consent prior to any study-specific procedures.
* Have adequate organ function.
* Have a performance status of less than or equal 1 on the Eastern Cooperative Oncology Group (ECOG).
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Prior radiation therapy for treatment of cancer is allowed to less than 25% of the bone marrow, and participants must have recovered from the acute toxic effects of their treatment prior to study enrollment. Prior radiation to the whole pelvis is not allowed.
* Males and females with reproductive potential: Must agree to use medically approved contraceptive precautions during the study and for 3 months following the last dose of study drug.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days of study enrollment, a clinical trial involving an investigational product or nonapproved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have moderate or severe cardiac disease:

  * Myocardial infarction within 6 months prior to study enrollment, unstable angina pectoris, New York Heart Association (NYHA) Class III/IV congestive heart failure, or uncontrolled hypertension.
  * Documented major electrocardiogram (ECG) abnormalities at the investigator's discretion.
  * Major abnormalities documented by echocardiography with Doppler.
  * Have significantly elevated brain natriuretic peptide (BNP) or elevated Troponin I at screening local laboratory tests.
  * Predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress.
  * Have a history of cardiac or aortic surgery.
* Have known positive tests for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C virus antibodies (HCVAbs).
* Have symptomatic central nervous system (CNS) malignancy or metastasis.
* Are unable to swallow tablets or capsules.
* Are pregnant or breastfeeding.
* Have serious preexisting medical conditions as follows:

  * Presence or history of interstitial pneumonitis.
  * Uncontrollable severe diabetes.
  * Presence of serious active infection or uncontrollable chronic infection.
  * Presence of liver cirrhosis with Child-Pugh Stage of B or C.
  * Other serious conditions judged by the investigator.
* Have previous or concurrent malignancy except for basal or squamous cell skin cancer (non-melanoma) and/or preinvasive carcinoma of the cervix, mucosal gastrointestinal or uterine carcinoma, or other solid tumors treated curatively and without evidence of recurrence for at least 3 years prior to enrollment.
* Have endocrine pancreatic tumors or ampullary cancer.
* Have current hematological malignancies.
* Have previously completed or withdrawn from this study or any other study investigating LY2157299.
* Have known allergies to LY2157299 or gemcitabine or any ingredient of LY2157299 or gemcitabine formulations.
* Are assessed as inadequate for the study by the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with LY2157299 Dose-Limiting Toxicities (DLT) | Cycle 1 (28 days)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of LY2157299 | Cycle 1: Predose on Day 1 through Day 28, Cycle 2 through last cycle: Predose on Day 1 (Cycle = 28 days; treatment estimated to last 4 cycles)
PK: Area Under the Plasma Concentration Versus Time Curve (AUC) of LY2157299 | Cycle 1: Predose on Day 1 through Day 28, Cycle 2 through last cycle: Predose on Day 1 (Cycle = 28 days; treatment estimated to last 4 cycles)
PK: Cmax of Gemcitabine | Cycle 1 (28 days): Predose on Day 8 through 2 hours after gemcitabine infusion on Day 8
PK: AUC of Gemcitabine | Cycle 1 (28 days): Predose on Day 8 through 2 hours after gemcitabine infusion on Day 8
Percentage of Participants with a Tumor Response | Baseline to study completion (estimated as 5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo